CLINICAL TRIAL: NCT04142788
Title: A Phase IV, Registry-based, Randomised, Controlled, Open-label Trial Investigating the Potential for Patiromer-facilitated Use of Higher Doses of MRAs in Addition to Standard Care to Improve Congestion, Well-being, Morbidity and Mortality
Brief Title: RELieving Increasing oEdema Due to Heart Failure
Acronym: RELIEHF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped due to low recruitment, which the Steering Committee and funder agreed could not be rectified.
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN17CA082; 2018-003662-14 (EudraCT Number)
Record Dates: First submitted 2019-10-08; First posted 2019-10-29 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure，Congestive
MeSH Terms: conditions — Heart Failure | interventions — patiromer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard dose MRA (No Intervention): Participants in this arm will have titration to guideline-recommended doses of MRA attempted.
- Patiromer and high dose MRA (Experimental): Participants assigned to patiromer may be titrated to 200mg/day spironolactone or the highest licensed dose of eplerenone (50mg/day).
  Interventions: Drug: Patiromer

INTERVENTIONS:
Drug: Patiromer — Patiromer (8.4g/day to 25.2g/day) and spironolactone (up to 200mg/day) or eplerenone (up to 50mg/day if spironolactone not acceptable). Treatments should be titrated to maintain serum potassium close to the target of 4.5mmol/L.
  Other Names: Veltassa
  Arms: Patiromer and high dose MRA

SUMMARY:
This trial will investigate the potential for patiromer-facilitated use of higher doses of mineralocorticoid antagonists in addition to standard care (compared to standard care alone) to improve congestion, well-being and mortality in people who have worsening congestion due to heart failure and hyperkalaemia.

DETAILED DESCRIPTION:
People with worsening congestive heart failure may benefit from treatment with higher doses of MRA if they are administered patiromer to treat or prevent hyperkalaemia.

Potential participants with worsening heart failure will be identified by their care teams and asked to participate in a research registry. If eligible, registry participants will be asked to take part in the RELIEHF randomised trial.

The randomised trial will investigate whether patiromer allows patients with worsening heart failure to be titrated to higher doses of MRA (predominantly spironolactone). Participants assigned to patiromer may be titrated to 200mg/day spironolactone or the highest licensed dose of eplerenone (50mg/day). Participants who are not assigned to patiromer should have titration to guideline-recommended doses of MRA attempted.

The registry and trial will take place in about 100 secondary care sites across the UK. At the end of the trial, participants will be followed through their electronic medical records via record linkage for up to 10 years

ELIGIBILITY:
Inclusion Criteria

A. For the Screening Log (no follow-up envisaged nor linkage to electronic medical records)

1. ≥18 years
2. Heart failure in the investigators opinion (new onset or decompensated chronic heart failure)
3. Planned to receive>80mg/day of furosemide or equivalent (IV, SC or oral) in the next 24 hours.
4. Worsening symptoms & signs of congestion in the prior 10 days requiring at least one of the following:

   1. hospitalisation
   2. administration of intravenous diuretics
   3. an increase in the dose of loop diuretic by at least 40mg/day of furosemide (or equivalent) to a total of at least 80mg/day of furosemide (or equivalent)
   4. addition of a thiazide diuretic to treatment with a loop diuretic

B. For the Consented Registry (with linkage to electronic medical records)

1. Fulfils the criteria for the screening log
2. Able and willing to provide written informed consent for registry participation

C. For Randomised Trial Run-in

1. Fulfils criteria for the consented registry
2. Clinical diagnosis of heart failure for at least 4 weeks
3. Congestion as shown by at least one of the following:

   1. Peripheral oedema
   2. Raised venous pressure
   3. Inferior vena cava diameter >20mm
4. Cardiac dysfunction documented by at least one of the following in the previous three years:

   1. A LVEF<50%or a report of moderate or severe left ventricular dysfunction
   2. Left atrial diameter >3.0cm/m2 (body surface area)
   3. Elevated BNP or NT-proBNP (BNP >150ng/L if in sinus rhythm or >450ng/L if not in sinus rhythm; NT-proBNP >500ng/L if in sinus rhythm and >1500ng/L if not in sinus rhythm)
5. Able and willing to provide written informed consent for the randomised trial

D. For Randomisation

1. Serum potassium >5.0mmol/L

   * Patients with a serum potassium >5.0mmol/L may be randomised immediately unless they have severe hyperkalaemia requiring, in the investigators opinion, intravenous treatment or a potassium binding agent.
   * Severe hyperkalaemia should be managed according to the UK Renal Association guidelines of 2014 (https://renal.org/wp-content/uploads/2017/06/hyperkalaemia-guideline-1.pdf). Participants may be reconsidered for the trial once such interventions are no longer considered necessary.
   * Patients with a serum potassium ≤5.0mmol/L should be initiated on spironolactone or have the dose increased up to 100mg/day and randomised only if serum potassium exceeds 5.0mmol/L. Those intolerant of or unwilling to take spironolactone should be offered eplerenone titrated to a maximum dose of 50mg/day.
   * A run-in period of up to 35 days is permitted (the run-in period will usually occur during hospitalisation or a course of day-care or intense management).
2. After ingestion of a test-dose of patiromer,

   1. the patient is willing to continue in the trial
   2. the investigator considers the patient can follow instructions on preparing patiromer

      Exclusion criteria

      A, For the Screening Log & Registry

      - None

      B. For the Randomised Trial
      1. eGFR <30ml/minute/1.73m2 (if clinically appropriate, the dose of other agents such as loop diuretics, ACE inhibitors, angiotensin receptor blockers, beta-blockers and sacubitril-valsartan may be adjusted to allow eGFR to increase)
      2. Systolic BP <90mmHg
      3. Uncorrected valve disease as the main cause of heart failure in the investigators opinion
      4. Hepatic encephalopathy or known severe liver disease
      5. Infection currently requiring intravenous antibiotics or temperature >38°C
      6. Myocardial ischaemia currently requiring intravenous therapy or coronary intervention in the previous 7 days
      7. Arrhythmia requiring urgent cardioversion or intravenous therapy
      8. Severe hyperkalaemia requiring, in the investigator's opinion, intravenous treatment or a potassium-binding agent
      9. The patient is already receiving a potassium-binding agent (this includes patiromer) or the treating physician has already decided to use one
      10. Known hypersensitivity to patiromer or any of the excipients
      11. Known intolerance to both spironolactone and eplerenone (not including hyperkalaemia)
      12. Known hypersensitivity to the active substance or excipients of spironolactone and eplerenone as per the current Summary of Product Characteristics (Note: actual medicine supplied to participants will vary depending on local arrangements)
      13. Women of childbearing potential. For the purposes of this trial this means any woman aged <60 years unless they have had a hysterectomy or bilateral tubal ligation or are aged >50 years and have undergone the menopause and had amenorrhea for at least 3 years
      14. Patients taking the following systemic medicines:

          * strong inhibitors of CYP 3A4 (e.g. itraconazole, ketoconazole, ritonavir, nelfinavir, clarithromycin, telithromycin and nefazodone)
          * Lithium
          * Tacrolimus or Cyclosporin
      15. The combination of an angiotensin converting enzyme (ACE) inhibitor and an angiotensin receptor blocker (ARB)
      16. Rare hereditary problems of galactose or fructose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
      17. Known amyloid heart disease
      18. Cancer likely to cause death or major disability within the next three years
      19. Patients requiring mechanical circulatory support and
      20. Patients who do not develop a serum potassium >5.0mmol/L despite receiving up to 100mg/day of spironolactone or 50mg/day of eplerenone during the run in phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Cleland, Principal Investigator — University of Glasgow
Locations (11):
- United Kingdom (11):
  - Glasgow Royal Infirmary, Glasgow, Strathclyde
  - Basildon University Hospital, Basildon
  - Blackpool Victoria Hospital, Blackpool
  - Princess of Wales Hospital, Bridgend
  - Royal Devon and Exeter Hospital, Exeter
  - Queen Elizabeth University Hospital, Glasgow
  - Castle Hill Hospital, Hull
  - Victoria Hospital, Kirkcaldy
  - Guy's and St Thomas's Hospital, London
  - King's College Hospital, London
  - St George's Hospital, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened across 12 sites between 13/03/2020 and 16/03/2022. The first participant to the registry was consented on 26/08/2020 and the last participant was consented to the registry on 17/03/2022. Participants to the trial that successfully completed run-in were randomised between 14/10/2021 and 16/03/2022.
Pre-assignment Details: 139 participants entered the registry but the trial was stopped because of low recruitment into the run-in phase (due, in part at least, the COVID pandemic), and because of the 19 patients who did enter the run-in phase, despite receiving up to spironolactone 100mg/day or eplerenone 50mg/day, only 4 patients developed a serum potassium >5.0 mmol/L, which was a requirement to enter the randomised phase of the trial.
Period: Overall Study
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Trial terminated prematurely | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Customized [Count of Participants; unit: Participants]
  Age group (years): <50 | 0 | 0 | 0
  Age group (years): 50-60 | 2 | 1 | 3
  Age group (years): >60 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 2 | 2 | 4
  Ethnicity: Mixed/Multiple ethnic groups | 0 | 0 | 0
  Ethnicity: Asian/Asian British | 0 | 0 | 0
  Ethnicity: Black/African/Caribbean/Black British | 0 | 0 | 0
  Ethnicity: Other ethnic group | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom: Scotland | 0 | 0 | 0
  United Kingdom: England | 0 | 2 | 2
  United Kingdom: Wales | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: "Congestion Index" on Day 60
Description: To find out whether administering patiromer and higher-dose MRA improves evidence of congestion on Day 60 compared to standard care.
Time Frame: After 400 patients have been evaluated at Day 60
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Morbidity/Mortality
Description: Composite of time to need for parenteral diuretic therapy (subsequent to initial discharge) for worsening or recalcitrant heart failure, (re-)hospitalisation for worsening heart failure or non-cancer deaths.
Time Frame: Through study completion
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Morbidity and Mortality
Description: Composite of time to (re-)hospitalisation or death
Time Frame: Periodically up to 10 years
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Dose of MRA
Description: Dose of MRA achieved for all trial participants
Time Frame: Days 7 and 60
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Congestion Index
Description: Congestion Index score for all trial participants
Time Frame: Days 7 and 60
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Days Dead or Hospitalised During the First 60 Days
Description: Days dead or hospitalised during the first 60 days for all trial participants
Time Frame: Through 60 days
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Quality of Life (EQ-5D)
Description: Quality of Life using validated EQ-5D questionnaire for all trial participants (visual analogue score - min 0, max 100, higher means better outcome; calculated score min 0, max 1, higher means better outcome)
Time Frame: Days 7 and 60
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Quality of Life Kansas City Cardiomyopathy Questionnaire (KCCQ-12)
Description: Quality of Life using validated KCCQ-12 questionnaire for all trial participants (score - min 0, max 100; higher means better outcome)
Time Frame: Days 7 and 60
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: NYHA Class
Description: NYHA class (I-IV) for all trial participants
Time Frame: Days 7 and 60
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Patient Global Assessment
Description: Patient Global Assessment to measure quality of life for all trial participants (ranges from markedly improved to markedly worsened; markedly improved means a better outcome)
Time Frame: Days 7 and 60
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Reduced All-cause Mortality
Description: All-cause mortality for all trial participants
Time Frame: Through study completion, up to 5 years
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Reduced Non-cancer Mortality
Description: Non-cancer mortality for all trial participants
Time Frame: Through study completion, up to 5 years
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Reduced Cardiovascular Mortality
Description: Cardiovascular mortality for all trial participants
Time Frame: Through study completion, up to 5 years
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Reduced Mortality/Morbidity - HF/Non-cancer
Description: Days lost to hospitalisation for heart failure or non-cancer deaths over 12 months for all trial participants
Time Frame: During first year
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Reduced Mortality/Morbidity - Any
Description: Days lost to any hospitalisation or any death over 12 months for all trial participants
Time Frame: During first year
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: QALY
Description: Quality adjusted life-years for duration of the trial for all trial participants
Time Frame: Through study completion, up to 5 years
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Proportion Alive and Well at 12 Months
Description: Proportion alive and well at 12 months (well-being defined by KCCQ-12 score) for all trial participants
Time Frame: At 12 months
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Dose of MRA
Description: Dose of MRA for all trial participants
Time Frame: At 6 months and 12 months
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Dose of Oral Diuretics Other Than MRA
Description: Dose of oral diuretics other than MRA for all trial participants
Time Frame: At 6 months and 12 months
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: NYHA Class
Description: NYHA class (I-IV) for all trial participants
Time Frame: At 6 months and 12 months
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Patient Global Assessment
Description: Patient Global Assessment to measure quality of life for all trial participants
Time Frame: At 6 months and 12 months
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Participant Characteristics and Assessment of Morbidity and Mortality
Description: Time to cardiovascular (re-)hospitalisation or non-cancer death for registry/trial participants
Time Frame: Periodically up to 10 years
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Participant Characteristics/Assessment of Morbidity/Mortality
Description: Time to heart failure (re-)hospitalisation or non-cancer death for registry/trial participants
Time Frame: Periodically up to 10 years
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Characteristics and Assessment of Morbidity/Mortality
Description: Incidence rate for hospitalisation for registry/trial participants
Time Frame: Periodically up to 10 years
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Characteristics/Assessment of Morbidity/Mortality
Description: Time to death (all-causes, cardiovascular causes, heart failure causes, cancer causes, and other) for registry and trial participants
Time Frame: Periodically up to 10 years
Population: Data were not collected due to early termination of the study.
Arm/Group | Standard Dose MRA | Patiromer and High Dose MRA
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 15 months due to early study termination
Description: Serious Adverse Event data were collected for all individuals entering run-in, regardless of whether or not they were subsequently randomised. Other [non-serious] adverse events were not collected as part of the study for the Run-in and Not Randomised Arm.
Groups:
- Run-in and Not Randomised: Participants with a serum potassium <=5.0mmol/L who are not currently receiving an MRA will first be given spironolactone (or eplerenone#) 25mg once daily and randomised to patiromer or not, if and when their serum potassium is >5.0mmol/L. If serum potassium does not exceed 5.0mmol/L within 72 hours, the dose of spironolactone may be increased to 50mg/day and after a further 72 hours to 100mg/day. Those intolerant of or unwilling to take spironolactone should be offered eplerenone (maximum dose 50mg/day).
  Participants with a serum potassium <=5.0mmol/L who are currently receiving an MRA at a dose of <50mg/day will be initiated on spironolactone 50mg once daily (or eplerenone#) or if currently already receiving 50mg/day, spironolactone 100mg/day (the maximum dose of eplerenone is 50mg/day). They will be randomised to receive patiromer or not, only once their serum potassium is >5.0mmol/L.
  [# only those intolerant of, or unwilling to take, spironolactone should be offered eplerenone]
Arm/Group | Run-in and Not Randomised | Standard Dose MRA | Patiromer and High Dose MRA
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in and Not Randomised (N=15) | Standard Dose MRA (N=2) | Patiromer and High Dose MRA (N=2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Cystoscopy (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Acute hyponatremia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in and Not Randomised (N=0) | Standard Dose MRA (N=2) | Patiromer and High Dose MRA (N=2)
Cardioversion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of the trial resulted in small numbers of patients recruited and no available analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT04142788/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT04142788/SAP_001.pdf